CLINICAL TRIAL: NCT06021067
Title: Dead Mesenchymal Stem Cells for the Treatment of Radiation Lung Injury
Brief Title: Dead Mesenchymal Stem Cells for Radiation Lung Injury
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RLI2023
Record Dates: First submitted 2023-06-24; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Radiation Lung Injury
Keywords: Dead Mesenchymal Stem Cells; Radiation Lung Injury; Treatment

STUDY DESIGN:
Intervention Model Description: one-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Death mesenchymal stem cell therapy plus standard treatment for radiation pneumonia (Experimental): Subjects (n=3) received a standard treatment regimen combined with a pre-specified starting dose of dead mesenchymal stem cells (2.0×10^7 for 60kg patient), infusion every 3 days, continuous infusion 4 times, treatment duration is 4~6 weeks. . If dose-limiting toxicity (DLT) does not occur within 30 days of the first administration, the dose is escalated by three times.
  Interventions: Biological: Death mesenchymal stem cell

INTERVENTIONS:
Biological: Death mesenchymal stem cell — A standard treatment regimen combined with a pre-specified starting dose of dead mesenchymal stem cells (2.0×10^7 for 60kg patient), infusion every 3 days, continuous infusion 4 times, treatment duration is 4~6 weeks.

SUMMARY:
The aim of this single center, single arm and prospective study is to explore the safety and efficacy of hDMSCs in the treatment of radiation pneumonitis.

DETAILED DESCRIPTION:
As a single-center, single-arm, prospective clinical trial, this study aims to explore the safety and efficacy of hDMSCs in the treatment of radiation pneumonia. This study will include patients who have received chest radiation therapy and are diagnosed with radiation lung injury based on clinical manifestations and changes in chest CT imaging. The degree of lung injury is graded according to CTCAE v5.0 criteria, and the corresponding standard treatment is received according to its grade. Using the 3+3 design for dose climbing, according to the order of patient inclusion, the first 3 patients (cohort 1) are treated with a standard treatment regimen combined with a pre-specified starting dose of dead mesenchymal stem cells (this study does not set up a live MSC group as a control). There are currently no relevant research results of previous human trials. The starting dose is obtained by our preclinical research. The mouse dose is 1×10^5/pc/30g, that is, the effective dose of mice is 3.3×10^6/kg. The dose of mice is 10 times that of humans, and the effective dose of humans is 3.3×10^5/kg. Therefore, the clinical effective dose of 60kg patients is 2.0×10^7, infusion every 3 days, continuous infusion 4 times, treatment duration of 4~6 weeks. During the dose-limited toxicity (DLT) observation period (30 days), observe the number of cases of DLT in 3 patients to determine whether to maintain the current dose group or adjust the dose group. If the dose of dead mesenchymal stem cells needs to be increased, the dose is ramped up by 3 times the starting dose (i.e., the second gradient dose is 6.0×10^7) until the number of patients in either dose group reaches 6 or the dose group adjustment is not possible. To determine the optimal therapeutic dose for the treatment of radiation lung injury using death mesenchymal stem cells in combination with standard therapy. A total of 15 patients were planned to be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Received chest radiotherapy;
* EOCG PS score of 0 to 3 points;
* Diagnosis of radiation lung injury by the attending physician, grade 2 to 3 (according to the CTCAE v5.0 standards);
* Main organs function is normal, that meet the following criteria: blood routine examination (within 7 days of unused hematopoietic growth factors and blood transfusion) : ANC ≥ 1.5 x 10^9 / L, PLT ≥ 80 x 10^9 / L, HGB ≥ 80 g/L;Biochemical examination: TBil ≤ 1.5 x ULN (upper limit of normal);ALT or AST ≤ 2.5 x ULN; Creatinine clearance ≥ 60 mL/min (Cockcroft - Gault formula); Blood coagulation function: INR or PT ≤ 1.5 x ULN, if the subjects are receiving anticoagulant therapy, as long as the scope of PT in anticoagulant drugs for it. Heart function examination, electrocardiogram (ECG) normal or abnormal ECG (by the researchers to determine the clinical significance). Heart doppler ultrasound assessment: LVEF ≥ 50%;
* Radiation lung injury lasts less than 2 months；
* Survival expectation ≥6 months;
* Signed and dated written informed consent

Exclusion Criteria:

* Pregnant or lactating women, men and women of childbearing age who are unwilling or unable to take effective contraceptive measures;
* People with a history of chronic bronchitis, emphysema, or cor pulmonale;
* History of lung resection surgery;
* Tumor progression;
* People with severe lung infection;
* Uncontrollable severe systemic diseases (e.g., central nervous system, cardiovascular system, blood system, digestive system, endocrine system, respiratory system, genitourinary system, immune system, etc.) and psychosis;
* Serious cardiovascular events: a period of 6 months in heart failure (NYHA class III level IV), myocardial infarction, unstable angina, severe arrhythmia, cerebral infarction, cerebral hemorrhage;
* Abnormal liver and kidney function: AST and ALT exceed the upper limit of normal by 2.5 times. Serum creatinine is greater than 1.5 mg/dl in men and 1.4 mg/dl in women;
* Co-infection with HIV, Treponema pallidum, tuberculosis, influenza virus, adenovirus and other respiratory infections;
* Hemorrhage or thrombosis, bleeding or anticoagulant drugs;
* Combined with cachexia or other organ failure (requiring organ support);
* Shock or invasive ventilation;
* Combined with pulmonary interstitial pneumonia caused by other reasons or damage, or lung imaging showed radioactive lung injury diagnosed with pulmonary interstitial pneumonia or damage before;
* Patients who have participated in clinical studies of stem cells;
* The investigators believed that there were other reasons why participants were not suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-09-10 (Estimated); Primary Completion 2024-09-10 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
The number of adverse events | up to 1 year
  The number of adverse events occurring within a given time frame will be reported according to CTCAE v5.0 to assess overall safety.

SECONDARY OUTCOMES:
Chest contrast-enhanced CT will be used to assess changes in lung injury after treatment | up to 1 year
  Chest contrast-enhanced CT will be performed at 1, 2, 3, 6, and 12 months after completion of dead mesenchymal stem cell injection, and the change in the proportion of total lesions to total lung volume will be calculated, i.e., (proportion of total lesions to total lung volume - proportion of total lesions to total lung volume at baseline) / proportion of total lesions to total lung volume at baseline.
Blood gas analysis will be performed after 1 month of dead mesenchymal stem cell injection. | up to 1 year
  At 1 month after completion of the injection of dead mesenchymal stem cells, changes in blood gas analysis will be observed to assess lung function.
Pulmonary function test will be performed after 1, 2, 3, 6, 12month of dead mesenchymal stem cell injection. | up to 1 year
  At after 1, 2, 3, 6, 12month completion of the injection of dead mesenchymal stem cells, pulmonary function test will be performed to assess recovery of lung function.
6-minute walking tests will be performed after 1, 2, 3, 6, 12month of dead mesenchymal stem cell injection. | up to 1 year
  At 1, 2, 3, 6 and 12 months after the completion of dead mesenchymal stem cell therapy, 6-minute walking tests will be performed to evaluate the recovery of the subjects' cardiopulmonary condition.
St. George's Respiratory Questionnaire will be completed to estimate the quality of life after 1, 2, 3, 6, 12month of dead mesenchymal stem cell injection. | up to 1 year
  At 1, 2, 3, 6 and 12 months after the completion of dead mesenchymal stem cell therapy, St. George's Respiratory Questionnaire will be completed to evaluate the subjects' quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen-Yu Ding, Prof, Principal Investigator — Sichuan University
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alfouzan AF. Radiation therapy in head and neck cancer. Saudi Med J. 2021 Mar;42(3):247-254. doi: 10.15537/smj.2021.42.3.20210660. PMID 33632902
- [Background] Bracci S, Valeriani M, Agolli L, De Sanctis V, Maurizi Enrici R, Osti MF. Renin-Angiotensin System Inhibitors Might Help to Reduce the Development of Symptomatic Radiation Pneumonitis After Stereotactic Body Radiotherapy for Lung Cancer. Clin Lung Cancer. 2016 May;17(3):189-97. doi: 10.1016/j.cllc.2015.08.007. Epub 2015 Aug 29. PMID 26427647
- [Background] Giuranno L, Ient J, De Ruysscher D, Vooijs MA. Radiation-Induced Lung Injury (RILI). Front Oncol. 2019 Sep 6;9:877. doi: 10.3389/fonc.2019.00877. eCollection 2019. PMID 31555602
- [Background] Chun SG, Hu C, Choy H, Komaki RU, Timmerman RD, Schild SE, Bogart JA, Dobelbower MC, Bosch W, Galvin JM, Kavadi VS, Narayan S, Iyengar P, Robinson CG, Wynn RB, Raben A, Augspurger ME, MacRae RM, Paulus R, Bradley JD. Impact of Intensity-Modulated Radiation Therapy Technique for Locally Advanced Non-Small-Cell Lung Cancer: A Secondary Analysis of the NRG Oncology RTOG 0617 Randomized Clinical Trial. J Clin Oncol. 2017 Jan;35(1):56-62. doi: 10.1200/JCO.2016.69.1378. Epub 2016 Oct 31. PMID 28034064
- [Background] Madan R, Benson R, Sharma DN, Julka PK, Rath GK. Radiation induced heart disease: Pathogenesis, management and review literature. J Egypt Natl Canc Inst. 2015 Dec;27(4):187-93. doi: 10.1016/j.jnci.2015.07.005. Epub 2015 Aug 18. PMID 26296945
- [Background] Palma DA, Olson R, Harrow S, Gaede S, Louie AV, Haasbeek C, Mulroy L, Lock M, Rodrigues GB, Yaremko BP, Schellenberg D, Ahmad B, Senthi S, Swaminath A, Kopek N, Liu M, Moore K, Currie S, Schlijper R, Bauman GS, Laba J, Qu XM, Warner A, Senan S. Stereotactic Ablative Radiotherapy for the Comprehensive Treatment of Oligometastatic Cancers: Long-Term Results of the SABR-COMET Phase II Randomized Trial. J Clin Oncol. 2020 Sep 1;38(25):2830-2838. doi: 10.1200/JCO.20.00818. Epub 2020 Jun 2. PMID 32484754
- [Background] Jain V, Berman AT. Radiation Pneumonitis: Old Problem, New Tricks. Cancers (Basel). 2018 Jul 3;10(7):222. doi: 10.3390/cancers10070222. PMID 29970850
- [Background] Maria OM, Maria AM, Ybarra N, Jeyaseelan K, Lee S, Perez J, Shalaby MY, Lehnert S, Faria S, Serban M, Seuntjens J, El Naqa I. Mesenchymal Stem Cells Adopt Lung Cell Phenotype in Normal and Radiation-induced Lung Injury Conditions. Appl Immunohistochem Mol Morphol. 2016 Apr;24(4):283-95. doi: 10.1097/PAI.0000000000000180. PMID 26200842
- [Background] Perez JR, Ybarra N, Chagnon F, Serban M, Lee S, Seuntjens J, Lesur O, El Naqa I. Tracking of Mesenchymal Stem Cells with Fluorescence Endomicroscopy Imaging in Radiotherapy-Induced Lung Injury. Sci Rep. 2017 Jan 19;7:40748. doi: 10.1038/srep40748. PMID 28102237
- [Background] Lee KC, Lin HC, Huang YH, Hung SC. Allo-transplantation of mesenchymal stem cells attenuates hepatic injury through IL1Ra dependent macrophage switch in a mouse model of liver disease. J Hepatol. 2015 Dec;63(6):1405-12. doi: 10.1016/j.jhep.2015.07.035. Epub 2015 Aug 11. PMID 26276675
- [Background] Islam D, Huang Y, Fanelli V, Delsedime L, Wu S, Khang J, Han B, Grassi A, Li M, Xu Y, Luo A, Wu J, Liu X, McKillop M, Medin J, Qiu H, Zhong N, Liu M, Laffey J, Li Y, Zhang H. Identification and Modulation of Microenvironment Is Crucial for Effective Mesenchymal Stromal Cell Therapy in Acute Lung Injury. Am J Respir Crit Care Med. 2019 May 15;199(10):1214-1224. doi: 10.1164/rccm.201802-0356OC. PMID 30521764
- [Background] Duan X, Lu L, Wang Y, Zhang F, Mao J, Cao M, Lin B, Zhang X, Shuai X, Shen J. The long-term fate of mesenchymal stem cells labeled with magnetic resonance imaging-visible polymersomes in cerebral ischemia. Int J Nanomedicine. 2017 Sep 8;12:6705-6719. doi: 10.2147/IJN.S146742. eCollection 2017. PMID 28932115
- [Background] Bruder SP, Jaiswal N, Ricalton NS, Mosca JD, Kraus KH, Kadiyala S. Mesenchymal stem cells in osteobiology and applied bone regeneration. Clin Orthop Relat Res. 1998 Oct;(355 Suppl):S247-56. doi: 10.1097/00003086-199810001-00025. PMID 9917644
- [Background] Zhou Y, Yamamoto Y, Xiao Z, Ochiya T. The Immunomodulatory Functions of Mesenchymal Stromal/Stem Cells Mediated via Paracrine Activity. J Clin Med. 2019 Jul 12;8(7):1025. doi: 10.3390/jcm8071025. PMID 31336889
- [Background] Song N, Scholtemeijer M, Shah K. Mesenchymal Stem Cell Immunomodulation: Mechanisms and Therapeutic Potential. Trends Pharmacol Sci. 2020 Sep;41(9):653-664. doi: 10.1016/j.tips.2020.06.009. Epub 2020 Jul 22. PMID 32709406
- [Background] Li L, Chen X, Wang WE, Zeng C. How to Improve the Survival of Transplanted Mesenchymal Stem Cell in Ischemic Heart? Stem Cells Int. 2016;2016:9682757. doi: 10.1155/2016/9682757. Epub 2015 Nov 22. PMID 26681958
- [Background] Sun T, Gao F, Li X, Cai Y, Bai M, Li F, Du L. A combination of ultrasound-targeted microbubble destruction with transplantation of bone marrow mesenchymal stem cells promotes recovery of acute liver injury. Stem Cell Res Ther. 2018 Dec 29;9(1):356. doi: 10.1186/s13287-018-1098-4. PMID 30594241
- [Background] Ramalho BDS, Almeida FM, Sales CM, de Lima S, Martinez AMB. Injection of bone marrow mesenchymal stem cells by intravenous or intraperitoneal routes is a viable alternative to spinal cord injury treatment in mice. Neural Regen Res. 2018 Jun;13(6):1046-1053. doi: 10.4103/1673-5374.233448. PMID 29926832
- [Background] He X, Hong W, Yang J, Lei H, Lu T, He C, Bi Z, Pan X, Liu Y, Dai L, Wang W, Huang C, Deng H, Wei X. Spontaneous apoptosis of cells in therapeutic stem cell preparation exert immunomodulatory effects through release of phosphatidylserine. Signal Transduct Target Ther. 2021 Jul 14;6(1):270. doi: 10.1038/s41392-021-00688-z. PMID 34262012
- [Background] Fadok VA, Bratton DL, Konowal A, Freed PW, Westcott JY, Henson PM. Macrophages that have ingested apoptotic cells in vitro inhibit proinflammatory cytokine production through autocrine/paracrine mechanisms involving TGF-beta, PGE2, and PAF. J Clin Invest. 1998 Feb 15;101(4):890-8. doi: 10.1172/JCI1112. PMID 9466984
- [Background] Ipseiz N, Uderhardt S, Scholtysek C, Steffen M, Schabbauer G, Bozec A, Schett G, Kronke G. The nuclear receptor Nr4a1 mediates anti-inflammatory effects of apoptotic cells. J Immunol. 2014 May 15;192(10):4852-8. doi: 10.4049/jimmunol.1303377. Epub 2014 Apr 16. PMID 24740500
- [Background] Chang CL, Leu S, Sung HC, Zhen YY, Cho CL, Chen A, Tsai TH, Chung SY, Chai HT, Sun CK, Yen CH, Yip HK. Impact of apoptotic adipose-derived mesenchymal stem cells on attenuating organ damage and reducing mortality in rat sepsis syndrome induced by cecal puncture and ligation. J Transl Med. 2012 Dec 7;10:244. doi: 10.1186/1479-5876-10-244. PMID 23217183
- [Background] Sung PH, Chang CL, Tsai TH, Chang LT, Leu S, Chen YL, Yang CC, Chua S, Yeh KH, Chai HT, Chang HW, Chen HH, Yip HK. Apoptotic adipose-derived mesenchymal stem cell therapy protects against lung and kidney injury in sepsis syndrome caused by cecal ligation puncture in rats. Stem Cell Res Ther. 2013;4(6):155. doi: 10.1186/scrt385. PMID 24451364
- [Background] Chen HH, Lin KC, Wallace CG, Chen YT, Yang CC, Leu S, Chen YC, Sun CK, Tsai TH, Chen YL, Chung SY, Chang CL, Yip HK. Additional benefit of combined therapy with melatonin and apoptotic adipose-derived mesenchymal stem cell against sepsis-induced kidney injury. J Pineal Res. 2014 Aug;57(1):16-32. doi: 10.1111/jpi.12140. Epub 2014 May 15. PMID 24761983
- [Background] Yip HK, Chang YC, Wallace CG, Chang LT, Tsai TH, Chen YL, Chang HW, Leu S, Zhen YY, Tsai CY, Yeh KH, Sun CK, Yen CH. Melatonin treatment improves adipose-derived mesenchymal stem cell therapy for acute lung ischemia-reperfusion injury. J Pineal Res. 2013 Mar;54(2):207-21. doi: 10.1111/jpi.12020. Epub 2012 Oct 30. PMID 23110436